CLINICAL TRIAL: NCT06564532
Title: Evaluating the Efficacy of a Marital Enhancement Application
Brief Title: Evaluative Conditioning and Relationship Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Principal Investigator, James McNulty, Principal Investigator, Florida State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: REL00000176
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Relationship, Marital

STUDY DESIGN:
Intervention Model Description: The investigators will recruit a sample of 500 active-duty servicemembers and their partners from Naval Medical Center at Portsmouth, VA. Half of all servicemembers will be randomly assigned to complete our EC procedure that pairs their partner with positive stimuli whereas the other half will be randomly assigned to complete a control procedure in which their partner is paired with neutral stimuli. Crossed with this manipulation, and also by random assignment, the partners of half the servicemembers will complete our EC procedure whereas the partners of the other half will complete the control procedure.
Who Masked: Participant
Masking Description: participants are not told the specific nature of the marital enhancement intervention and both experimental and control participants complete the same procedure with only one exception--whether their partner is paired with positive or neutral words and images.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Servicemember and partner paired with positive stimuli (Experimental): Both the servicemember and the partner of the servicemember see their partner paired with positive stimuli
  Interventions: Behavioral: Evaluatively conditioning participant to like partner; Behavioral: Evaluatively conditioning partner to like participant
- Servicemember partner paired with positive stimuli, servicemember paired with neutral stimuli (Experimental): The servicemember sees the partner paired with positive stimuli and the partner sees the servicemember paired with neutral stimuli
  Interventions: Behavioral: Evaluatively conditioning participant to like partner
- Servicemember partner paired with neutral stimuli, servicemember paired with positive stimuli (Experimental): The servicemember sees the partner paired with neutral stimuli and the partner sees the servicemember paired with positive stimuli
  Interventions: Behavioral: Evaluatively conditioning partner to like participant
- Servicemember and partner paired with neutral stimuli (No Intervention): Both the servicemember and the partner of the servicemember see their partner paired with neutral stimuli

INTERVENTIONS:
Behavioral: Evaluatively conditioning participant to like partner — The intervention is a computerized learning task that leads the participant to associate the partner with positive stimuli
  Arms: Servicemember and partner paired with positive stimuli; Servicemember partner paired with positive stimuli, servicemember paired with neutral stimuli
Behavioral: Evaluatively conditioning partner to like participant — The intervention is a computerized learning task that leads the partner to associate the participant with positive stimuli
  Arms: Servicemember and partner paired with positive stimuli; Servicemember partner paired with neutral stimuli, servicemember paired with positive stimuli

SUMMARY:
The overall objective is to evaluate the efficacy of a novel computerized learning procedure to enhance marital well-being among military members and their partners.

DETAILED DESCRIPTION:
Large bodies of research indicate that people's health, occupational performance, and job satisfaction depend critically on their marital well-being. Nevertheless, several challenges associated with military service, such as increased stress and physical separation from one's partner, can threaten marital well-being. Prior research by our team highlights the important marital implications of automatic partner attitudes, or the immediate affective reactions experienced when thinking about or interacting with one's partner. Most couples strengthen these partner attitudes through enjoyable experiences together, but servicemembers who are separated from their partners must forego such activities, and job-related stress can minimize the positivity of any joint activities that do occur. Evaluative Conditioning (EC) offers a way to strengthen automatic partner attitudes without direct experience with the partner through simple pairings of photos of the partner with positive words and images. Our pilot study of civilian couples demonstrated that couples randomly assigned to view photos of their partners paired with positive stimuli for 6-7 minutes every three days for six weeks experienced enhanced automatic partner attitudes and thus marital satisfaction over eight weeks relative to control couples.

The proposed research would use a RCT to test (a) the feasibility and efficacy of EC procedure among active duty servicemembers and (b) whether there is an additional benefit to having the partner also complete the EC procedure. Regarding the first objective, the investigators predict that people who view their partner paired with positive stimuli will demonstrate enhanced automatic partner attitudes and therefore higher levels of marital satisfaction and more positive relationship behaviors relative to people who view their partner paired with neutral stimuli. Regarding the second objective, the investigators expect that EC will be more effective when the partner also completes it, though the investigators suspect it will be effective even among servicemembers whose partners do not complete the procedure.

The aim of the proposed research is to conduct an RCT to determine (a) whether evaluative conditioning can enhance automatic partner attitudes and thereby marital satisfaction and behavior in a sample of active duty servicemembers and (b) whether any benefits of EC depend on whether one or both members of the couple complete the procedure.

The investigators will recruit a sample of 500 active-duty servicemembers and their partners from Naval Medical Center at Portsmouth, VA. Half of all servicemembers will be randomly assigned to complete our EC procedure that pairs their partner with positive stimuli whereas the other half will be randomly assigned to complete a control procedure in which their partner is paired with neutral stimuli. Crossed with this manipulation, and also by random assignment, the partners of half the servicemembers will complete our EC procedure whereas the partners of the other half will complete the control procedure. Both members of the couple will complete assessments of automatic partner attitudes and marital satisfaction at baseline and then again every two weeks for eight weeks. Couples will also engage in recorded marital discussions at baseline and the 8-week follow-up to assess behavior.

ELIGIBILITY:
Inclusion Criteria:

* one member of the couple is active-duty US military
* couple is married
* both couple members are at least 18 years old
* both couple members are proficient readers and speakers of English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Partner Evaluative Priming Procedure (McNulty et al., 2013) | Every two weeks for eight weeks
  Modeled after the evaluative priming task developed by Fazio et al. (1995), the task implicitly measures participants' automatically activated partner attitudes by measuring RTs to positive and negative words following exposure to primes of the partner. Primes will be photos primes of the partner appearing in one of four orientations in each photo: (a) a frontal view of the face, (b) a profile view of the face, (c) a frontal view of the entire body while standing, and (d) a frontal view of the entire body while sitting.
Couples Satisfaction Index (Funk & Rogge, 2007) | Every two weeks for eight weeks
  Questionnaire to assess self-reported satisfaction with the relationship
Verbal Tactics Coding Scheme (Sillars, 1982) | Eight weeks
  Qualitative coding scheme designed to identify direct and indirect oppositional statements during problem-solving discussions
Suicidality subscale of the Depressive Symptom Index (Metalsky & Joiner, 1997 | Every two weeks for eight weeks
  a well-validated measure that assesses the fre- quency and controllability of suicidal thoughts as agreement with four sets of four statements that increase in severity

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT06564532/ICF_000.pdf